CLINICAL TRIAL: NCT01541293
Title: Intrauterine Lidocaine for Pain Control During Laminaria Insertion Prior to Dilation & Evacuation (D&E)
Brief Title: Intrauterine Lidocaine for Laminaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-1928
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2013-10

CONDITIONS: Abortion, Induced; Pain Management
Keywords: Abortion, Induced; Laminaria; Pain management; Cervical preparation; Dilation and Evacuation
MeSH Terms: conditions — Agnosia; Dilatation, Pathologic | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrauterine Lidocaine (Experimental): The experimental arm will receive 100mg lidocaine (5mL of 2% concentration) instilled into the uterine cavity via a flexible trans-cervical catheter immediately prior to laminaria insertion.
  Interventions: Drug: Lidocaine
- Intrauterine Saline (Placebo Comparator): Placebo arm will receive 5mL of normal saline instilled into the uterine cavity via a flexible trans-cervical catheter immediately prior to laminaria insertion.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Lidocaine — 100mg of liquid lidocaine, single dose, instilled into the uterine cavity via a flexible trans-cervical catheter immediately prior to laminaria insertion.
  Arms: Intrauterine Lidocaine
Drug: Normal Saline — 5mL of normal saline, instilled into the uterus via a flexible trans-cervical catheter immediately prior to laminaria insertion.
  Arms: Intrauterine Saline

SUMMARY:
This is a study to investigate whether instilling a small amount of liquid lidocaine into the uterus will decrease pain felt by women during laminaria insertions done for cervical dilation prior to second trimester abortion.

The investigators hypothesize that women who receive intrauterine lidocaine in addition to a paracervical block will experience less pain than women who receive only a paracervical block.

ELIGIBILITY:
Inclusion Criteria:

* Can sign informed consent
* Healthy pregnant females
* Weight over 45kg
* Seeking abortion by dilation and evacuation in the second trimester of pregnancy
* Gestational age 14-24 weeks confirmed by clinic ultrasound

Exclusion Criteria:

* Known allergy or previous reaction to lidocaine, bupivicaine or other anesthetic agent
* Known allergy or previous reaction to ibuprofen or other NSAID

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Patient self-report of pain score during laminaria insertion, scored on a 100mm Visual Analog Scale | Immediately following laminaria insertion

SECONDARY OUTCOMES:
Patient self-report of maximum recalled pain during interval between laminaria insertion and abortion procedure, scored on a 100mm Visual Analog Scale | 24-48 hours after laminaria insertion

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Mercier, MD MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Mercier RJ, Liberty A. Intrauterine lidocaine for pain control during laminaria insertion: a randomized controlled trial. Contraception. 2014 Dec;90(6):594-600. doi: 10.1016/j.contraception.2014.07.008. Epub 2014 Jul 23. PMID 25139724